CLINICAL TRIAL: NCT01641731
Title: Efficacy and Safety of Specific Oral Tolerance Induction in Children Allergic to Cow's Milk Proteins According to Their Serum Specific IgE Level
Brief Title: Specific Oral Tolerance Induction in Children Allergic to Cow's Milk Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOTI_CMA_HULP
Record Dates: First submitted 2012-05-28; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Cow's Milk Protein Sensitivity
Keywords: cow's milk protein allergy; oral tolerance induction
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cow's milk (Active Comparator)
  Interventions: Other: Cow's milk
- Control group (No Intervention)

INTERVENTIONS:
Other: Cow's milk — Group I: Increase 2 mL until 10 mL, 10 mL until 50 mL, 20 mL until 100 mL and 50 mL until 200 mL was reached.
  Groups II and III: Doubling dose until 1 mL, increase 2 mL until 20 mL, 5 mL until 50 mL, 10 mL until 100 mL and 20 mL until 200 mL was reached.
  Arms: Cow's milk

SUMMARY:
Induction of oral tolerance in children allergic to cow's milk proteins is not risk-free. The analysis of factors that may influence the outcome is of utmost importance.

The aim of the study is to analyse the efficacy and safety of the induction phase of oral tolerance induction according to specific IgE level, as well as adverse events during the maintenance phase.

Patients allergic to cow's milk are to be included in an oral tolerance induction protocol. Patients will be grouped according to specific IgE levels in serum (ImmunoCAP) into group I (sIgE<3.5 kU/L), II (sIgE 3.5-17 kU/L) and III (>17-50kU/L). Allergic children with similar characteristics will included as a control group. Visits are established at 1, 6 and 12 months after the induction phase. Serum specific IgE levels to cow's milk and its proteins will be determined at inclusion, and at 6 and 12 months visits after the induction phase.

DETAILED DESCRIPTION:
Children allergic to cow's milk proteins (CMA) will be included. They have to be diagnosed with CMA during the first year of life and have attended periodic follow-up visits to our Allergy Clinic at Hospital La Paz (Madrid, Spain). Clinical data on personal history of asthma, allergy to other foods and positive reactions upon cow's milk ingestion along with their evolution from initial diagnosis will be recorded.

Prior to inclusion in the SOTI protocol, determination of serum specific IgE to cow's milk (CM), ALA, BLG and casein (ImmunoCAP, Phadia, Uppsala, Sweden) will be performed and current clinical status will be confirmed by oral food challenge (OFC) with cow's milk. An open OFC with CM (3 g of proteins per 100 mL) will be performed following a modified protocol according to the level of allergic sensitisation. Group I will start at a dose of 2 mL, and those in groups II and III started at a dose of 0.005 mL. In both protocols doses will be doubled until objective clinical reactivity is achieved.

Determination of serum specific IgE to cow's milk and its proteins will be performed in the follow-up at 6 and 12 months visits.

In order to evaluate the influence of the level of sensitisation in the result of SOTI, patients will be classified into three groups according to the level of sIgE for CM and/or its proteins: group I (0.35-3.5 kU/L, CAP Class I and II); group II (>3.5-17 kU/L, CAP Class III); group III (>17-50kU/L, CAP Class IV). The highest sIgE level against any of the CM or its proteins will determine the group of inclusion.

A control group of cow's milk allergic children, with similar levels of sIgE, will be included in order to evaluate the natural evolution to tolerance in CMA. They will be followed for one year, after which, clinical reactivity with OFC will be again confirmed. These control patients will selected among those who, after the initial OFC, refuse to undergo SOTI.

Specific Oral Tolerance Induction:

The initial dose for SOTI will be the previous dose that elicited symptoms in the OFC. Group I doses will be upped weekly in the hospital setting, and patients will maintain that dose twice daily at home. Groups II and III also will start with the previous dose that elicited symptoms in the OFC, but will receive incremental doses daily in the hospital setting until they reach a dose of 1 mL. Achieving an intake of 200 mL of milk (6 g of proteins) twice a day, which is the usual amount for patients of that age, will be considered complete tolerance.

Reactions occurring during the induction phase at the hospital will be treated according to the severity of symptoms. If patients present with mild non-objective symptoms, the same dose will be repeated. If the reaction is objective and limited to local symptoms, the previous dose will be given after the resolution of symptoms. If the reaction is generalised, involving two organ systems, SOTI will be continued with a dose which is two doses previous to the one that elicited symptoms. If the reaction involves three organ systems, the next dose administered will be reduced three steps in the dosage protocol. Written instructions will be given to parents regarding how to treat possible adverse reactions at home.

After the induction phase, patients will continue to consume 200 mL milk twice daily and dairy products were allowed freely.

In the maintenance phase, follow-up visits are scheduled at one month, six months and one year after finishing the induction phase. Data on tolerance of cow's milk and dairy products will be recorded. Adverse events upon ingestion will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

-Patients diagnosed with cow's milk allergy meeting the following criteria: Immediate-type clinical manifestations, skin (urticaria, angioedema and/or erythema), digestive (acute vomiting and/or diarrhea) or respiratory (bronchospasm and/or rhinitis) involvement in the first two hours after cow's milk ingestion.

Skin test readings ≥ 3 mm and specific IgE titers > 0.35 kU/l for whole cow's milk or someone of isolated CMPs (casein, alpha-lactalbumin, beta-lactoglobulin )

* Age 4 years old or older
* Specific IgE (measured by ImmunoCAP) lower than 50 KU/L for cow's milk or its proteins
* Positive oral food challenge with a dose higher than 2 mL
* Written informed consent signed by parents or legal representatives

Exclusion Criteria:

* Age younger than 4 y.o.
* Specific IgE higher than 50 kU/L
* Patients in whom oral food challenges is contraindicated, because of having a positive accidental reaction with moderate or severe symptoms in the previous 12 months prior to the inclusion.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Tolerance to cow's milk | 12 months
  After administration of 250ml of milk, the patient is evaluated to determined if the milk is tolerated or not.

SECONDARY OUTCOMES:
Adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen García-Ara, MD, PhD, Principal Investigator — Instituto de Investigación Sanitaria Hospital Universitario La Paz
Locations (1):
- Servicio de Alergia Infantil, Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Background] Longo G, Barbi E, Berti I, Meneghetti R, Pittalis A, Ronfani L, Ventura A. Specific oral tolerance induction in children with very severe cow's milk-induced reactions. J Allergy Clin Immunol. 2008 Feb;121(2):343-7. doi: 10.1016/j.jaci.2007.10.029. Epub 2007 Dec 26. PMID 18158176
- [Background] Zapatero L, Alonso E, Fuentes V, Martinez MI. Oral desensitization in children with cow's milk allergy. J Investig Allergol Clin Immunol. 2008;18(5):389-96. PMID 18973104
- [Background] Caminiti L, Passalacqua G, Barberi S, Vita D, Barberio G, De Luca R, Pajno GB. A new protocol for specific oral tolerance induction in children with IgE-mediated cow's milk allergy. Allergy Asthma Proc. 2009 Jul-Aug;30(4):443-8. doi: 10.2500/aap.2009.30.3221. Epub 2009 Mar 13. PMID 19288980
- [Background] Staden U, Rolinck-Werninghaus C, Brewe F, Wahn U, Niggemann B, Beyer K. Specific oral tolerance induction in food allergy in children: efficacy and clinical patterns of reaction. Allergy. 2007 Nov;62(11):1261-9. doi: 10.1111/j.1398-9995.2007.01501.x. PMID 17919140
- [Background] Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG, Matsui EC, Burks AW, Wood RA. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol. 2008 Dec;122(6):1154-60. doi: 10.1016/j.jaci.2008.09.030. Epub 2008 Oct 25. PMID 18951617
- [Derived] Garcia-Ara C, Pedrosa M, Belver MT, Martin-Munoz MF, Quirce S, Boyano-Martinez T. Efficacy and safety of oral desensitization in children with cow's milk allergy according to their serum specific IgE level. Ann Allergy Asthma Immunol. 2013 Apr;110(4):290-4. doi: 10.1016/j.anai.2013.01.013. Epub 2013 Feb 14. PMID 23535095